CLINICAL TRIAL: NCT03769688
Title: VMT-01: Safety and Efficacy of Vaginal Microbiota Transplant (VMT) in Women With Bacterial Vaginosis (BV)
Brief Title: Safety and Efficacy of Vaginal Microbiota Transplant (VMT) in Women With Bacterial Vaginosis (BV)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Replaced with different study at another site.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00090758
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; cervicovaginal secretions; vaginal microbiota
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Early Detection of Cancer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cervicovaginal secretions (Experimental): Participants will receive standard of care antibiotics (vaginal Metronidazole gel). After standard antibiotic treatment, participants will receive a single intravaginal dose of cervicovaginal secretions (10 mg in 1 ml total volume, 0.9 ml normal saline).
  Interventions: Drug: Cervicovaginal secretions; Drug: Metronidazole gel; Diagnostic Test: Screening tests; Behavioral: Activities restriction
- Saline placebo (Placebo Comparator): Participants will receive standard of care antibiotics (vaginal Metronidazole gel). After standard antibiotic treatment, participants will receive a single intravaginal dose of sterile saline placebo (1 ml total volume).
  Interventions: Drug: Metronidazole gel; Diagnostic Test: Screening tests; Behavioral: Activities restriction; Other: Sterile Saline placebo

INTERVENTIONS:
Drug: Cervicovaginal secretions — Same as arm descriptions
  Arms: Cervicovaginal secretions
Drug: Metronidazole gel — 5 day course of vaginal MetroGel will be used prior to VMT intervention.
Diagnostic Test: Screening tests — Diagnostic testing for a broad range of infectious pathogens in blood, vaginal swab, and urine samples, for general immunocompetence, and for potential pregnancy.
Behavioral: Activities restriction — Required abstinence from sexual intercourse, usage of insertive vaginal feminine products (i.e. Tampons, menstrual cups, sex toys), other vaginal products (cleansing products, spermicides, lubricants, hygiene powders and sprays), and avoidance of behaviors including taking baths, going swimming, sitting in hot tub, or wearing thong underwear. Sanitary napkins are acceptable.
Other: Sterile Saline placebo — This will be administered as a placebo in place of cervicovaginal secretions
  Arms: Saline placebo

SUMMARY:
The composition of a woman's vaginal microbiota has a significant impact on her reproductive tract health and general quality of life. Approximately one-third of all women currently have bacterial vaginosis (BV), a polymicrobial condition in which the vaginal microbiota is not dominated by Lactobacillus species, leading to increased risk of various reproductive tract maladies and negative impact on well-being. It has been suggested by epidemiological studies that vaginal microbiota are readily transferable from one woman to another. Here, investigators aim to explore the hypothesis that vaginal microbiota can be engrafted from one woman to another in a controlled clinical setting by using cervicovaginal secretions (CVS), a process referred to as vaginal microbiota transplant (VMT).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria that apply to potential Donor participants:

1. Capable of reading and writing English and voluntarily provide written informed consent to participate in the study and comply with all study procedures.
2. Generally healthy, pre-menopausal women age 18-45 years old.
3. Regular predictable menstrual cycles or amenorrheic for at least 3 months due to use of long-acting progestin or continuous use of oral contraceptives.
4. Free of vaginal symptoms, such as odor, discharge, or itching.
5. Willing to be asked questions about personal medical, sexual, and behavioral history.
6. Willing to self-collect cervicovaginal secretions and vaginal swab samples.
7. Agree to abstain from using insertive vaginal feminine products (i.e. Tampons, menstrual cups, sex toys), other vaginal products (cleansing products, spermicides, lubricants, hygiene powders and sprays), vaginal and anal intercourse, taking baths, going swimming, sitting in hot tub, or wearing thong underwear during the entire sample donation period (from screening to the final donation). Sanitary napkins are acceptable.

Inclusion criteria that apply to potential Recipient participants:

1. Capable of reading and writing English and voluntarily provide written informed consent to participate in the study and comply with all study procedures.
2. Generally healthy, pre-menopausal women age 18-45 years old.
3. Experiences recurrent bacterial vaginosis (BV) (at least 3 diagnoses in their lifetime), and has received treatment for BV on at least 1 prior occasion in the past 5 years.
4. Currently needing treatment for vaginal symptoms clinically diagnosed as BV (>= 3 Amsel criteria and confirmed in the laboratory by Nugent score >= 4) and suitable for 0.75% metronidazole vaginal antibiotic treatment.
5. Regular predictable menstrual cycles or amenorrheic for at least 3 months due to use of long-acting progestin or continuous use of oral contraceptives.
6. Women who are not sterilized or who are not using an Intra-uterine Device (IUD) or form of hormonal contraception must agree to barrier contraception (i.e. Condoms, diaphragm) for heterosexual intercourse during the study. Counseling will be provided for use of barrier contraception without the use of adjunctive spermicide or lubricant.
7. Willing to be asked questions about personal medical, sexual, and behavioral history.
8. Willing to self-collect cervicovaginal secretions and vaginal swab samples.
9. Willing to undergo VMT procedure.
10. Agree to abstain from vaginal intercourse, unless using a condom, for at least the 28 days after the VMT procedure. Condoms will be provided.
11. Agree to avoid taking baths, swimming, sitting in a hot tub, or wearing thong underwear for at least the 28 days after the VMT procedure.
12. Agree to abstain from using insertive vaginal feminine products (i.e. Tampons, menstrual cups, sex toys), vaginal cleansing products, spermicides, lubricants, or other vaginal products not approved by the study investigators after the VMT procedure through visit 8 (~6 months). Sanitary napkins are acceptable.

Exclusion Criteria:

Exclusion criteria that apply to potential Donor participants:

1. Any history of bacterial vaginosis, recurrent yeast infection, trichomoniasis, syphilis, human papilloma virus (HPV) including genital warts, high grade pap smear, herpes, pelvic inflammatory disease, recurrent urinary tract infection, mycoplasma.
2. Testing positive for HIV, Hepatitis A/B/C, syphilis, Human T-lymphotrophic Virus (HTLV)-I/II, WNV, Epstein-Barr Virus (EBV), rubella, toxoplasma gondii, Herpes Simplex Virus (HSV)-1/2, yeast or bacteria that are considered pathogenic/abnormal and/or show antibiotic resistance, chlamydia, gonorrhea, mycoplasma genitalium, trichomonas vaginalis, HPV.
3. Cervicovaginal secretions (CVS) not dominated by one of the common vaginal lactobacillus species, as determined by qPCR.
4. Currently pregnant or breastfeeding.
5. History of gonorrhea or chlamydia within 12 months prior to screening.
6. Travel or sexual partner travel to regions or countries where Ebola or Zika outbreaks occurred in the past 12 months.
7. Any other medical, travel, or behavioral history that deems donors of human cells, tissues, and cellular and tissue-based products (HCT/Ps) ineligible.
8. HIV/AIDS or other immunodeficiency, or testing out of the range of normal clinical parameters for general measures of immunocompetence.
9. Hysterectomy.
10. Use of vaginal ring (e.g., NuvaRing) within 3 days of screening or during the course of the study.
11. Investigational drug use within 30 days or 10 half-lives of the drug, whichever is longer, of enrollment visit, or planned participation in an investigational drug study while participating in this study.
12. IUD insertion or removal, cervical cryotherapy, or cervical laser treatment within 2 months prior to screening.
13. Any condition requiring regular periodic use of systemic antibiotics during the study.
14. New use of long-acting hormonal treatments. Participant may be enrolled if stable (>3 months) or existing therapy as determined by the investigator.
15. Any social, medical, or psychiatric condition, including history of drug or alcohol abuse that in the opinion of the investigator would make it unlikely for the participant to comply with the study or would complicate interpretation of data from her participation.
16. Menopause defined as more than 12 consecutive months of amenorrhea without another known cause.
17. Irregular menstrual cycles that preclude scheduling appointments to avoid menstruation.
18. Donors will be screened for cytomegalovirus (CMV), Rubella, and Varicella Zoster Virus (VZV) IgG, which will not be a criterion for exclusion, but samples from CMV positive and/or Rubella positive and/or VZV positive Donors will only be matched with CMV positive and/or Rubella and/or VZV positive Recipients.
19. Abnormal finding on exam, which, in the opinion of the investigator, precludes participation.
20. Sexual history or current sexual behavior, or having sexual partners that engage in such behaviors, which introduces increased risk of sexually transmitted infections or exposure to pathogenic organisms.
21. Medication use, recent vaccinations, sources of income, or other behaviors, which in the opinion of the investigator, precludes participation.

Exclusion Criteria that apply to potential Recipient participants

1. Current pregnancy, within 2 months of pregnancy, planning to become pregnant within the next 6 months, and/or currently breastfeeding.
2. HIV/AIDS or other immunodeficiency.
3. Testing positive for HIV, HTLV-I/II, yeast infection, chlamydia, gonorrhea, mycoplasma genitalium, trichomonas, antibiotic-resistant bacteria in culture, or human Chorionic Gonadotrophin (hCG) (urine).
4. Hysterectomy.
5. High grade pap smear within the past year.
6. Use of vaginal ring (e.g., NuvaRing) during the course of the study.
7. Investigational drug use within 30 days or 10 half-lives of the drug, whichever is longer, of enrollment visit, or planned participation in an investigational drug study while participating in this study.
8. IUD insertion or removal, cervical cryotherapy, or cervical laser treatment within 2 months prior to screening.
9. Any condition requiring regular periodic use of systemic antibiotics during the study.
10. New use of long-acting hormonal treatments. Participant may be enrolled if stable (>3 months) or existing therapy as determined by the investigator.
11. Any social, medical, or psychiatric condition, including history of drug or alcohol abuse that in the opinion of the investigator would make it unlikely for the participant to comply with the study or would complicate interpretation of data from her participation.
12. Menopause defined as more than 12 consecutive months of amenorrhea without another known cause.
13. Recipients will be screened for cytomegalovirus (CMV), Rubella, and Varicella Zoster Virus (VZV) IgG, which will not be a criterion for exclusion, but samples from CMV positive and/or Rubella positive and/or VZV positive Donors will only be matched with CMV positive and/or Rubella and/or VZV positive Recipients.
14. Abnormal finding on exam, which, in the opinion of the investigator, precludes participation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Bacteria engraftment as assessed by ribosomal (rDNA) gene sequencing | 28 days
  Detection of Donor vaginal Lactobacillus in Recipient by 16S rDNA gene sequencing (~1% or greater relative abundance by read count)

SECONDARY OUTCOMES:
Bacteria engraftment as assessed by rDNA gene sequencing | 10 days
  Detection of Donor vaginal Lactobacillus in Recipient by 16S rDNA gene sequencing (~1% or greater relative abundance by read count)
Bacterial communities as assessed by rDNA gene sequencing | At screening , and then follow-up (~7 months)
  Identify bacterial communities colonizing the vagina at screening in women with bacterial vaginosis and after antibiotic and CVS treatment by 16S rDNA sequencing
Bacterial vaginosis recurrence as assessed by Amsel's criteria | Up to 6 months after VMT procedure
  Determination of recurrence of BV in participants by Amsel's criteria. Amsel's criteria includes the presence of a homogeneous vaginal discharge, pH of the vagina being > 4.5, the presence of clue cells in gram stained vaginal discharge smears and a positive whiff test. According to Amsel, if 3 of the 4 criteria are positive, the patient has bacterial vaginosis
Bacterial vaginosis recurrence as assessed by Nugent score | Up to 6 months after VMT procedure
  Determination of recurrence of BV in participants by Nugent score. The Nugent score is calculated by assessing for the presence of large Gram-positive rods (Lactobacillus morphotypes; decrease in Lactobacillus scored as 0 to 4), small Gram-variable rods (Gardnerella vaginalis morphotypes; scored as 0 to 4), and curved Gram-variable rods (Mobiluncus spp. morphotypes; scored as 0 to 2). A total score of 7 to 10 is consistent with bacterial vaginosis without culture.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ensign, PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No